CLINICAL TRIAL: NCT07100873
Title: A Phase 1 Study of ADI-001 Anti-CD20 CAR-engineered Allogeneic Gamma-Delta (γδ) T Cells in Adults With Treatment-refractory Rheumatoid Arthritis
Brief Title: A Phase 1 Study of ADI-001 in Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adicet Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADI-001-106
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Experimental: Run-in (Experimental)
  Interventions: Drug: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide
- Experimental: Part 1a (Experimental): Cy/Flu LD
  Interventions: Drug: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide
- Experimental: Part 1b (Experimental): Cy-only LD
  Interventions: Drug: ADI-001; Drug: Cyclophosphamide
- Experimental: Part 2a (Experimental): Cy/Flu LD
  Interventions: Drug: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide
- Experimental: Part 2b (Experimental): Cy-only LD
  Interventions: Drug: ADI-001; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: ADI-001 — Anti-CD20 CAR-T
Drug: Fludarabine — Chemotherapy for Lymphodepletion
  Arms: Experimental: Part 1a; Experimental: Part 2a; Experimental: Run-in
Drug: Cyclophosphamide — Chemotherapy for Lymphodepletion

SUMMARY:
ADI-001-106 is a phase 1 study of ADI-001 with a randomized, single-blind, parallel group design to compare two different LD regimens in subjects with treatment-refractory RA. The study will consist of different periods including screening, LD, treatment, and follow-up

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Fulfills the 2010 ACR-EULAR RA classification criteria
3. Agreement not to take traditional medicines and medications not prescribed by a doctor
4. Adequate hematological, liver, cardiac and pulmonary function

Exclusion Criteria:

1. Presence of severe liver disease, Child-Pugh class B or C.
2. Autoimmune disease requiring prednisone higher than 0.5 mg/kg/day (or corticosteroid equivalent).
3. Subjects unwilling to participate in an extended safety monitoring period (LTFU protocol)
4. History of a clinically significant infection (including sepsis, pneumonia, bacteremia, fungal, viral and opportunistic infections) within 4 weeks prior to first dose of study drug which in the opinion of the Investigator may compromise the safety of the subject in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Subjects with Dose Limiting Toxicities within each dose level cohort | 28 days
  This primary endpoint will be used to evaluate safety and tolerability of AD1-001 in subjects with treatment-refractory RA

CONTACTS AND LOCATIONS:
Locations (1):
- Adicet Clinical Trials, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No